CLINICAL TRIAL: NCT01218971
Title: A Multicenter Double-Blind Extension of Alkermes Study ALK21-003 to Evaluate the Long-Term Safety of Medisorb® Naltrexone
Brief Title: ALK21-003EXT: An Extension of Study ALK21-003 (NCT01218958) to Test the Long-term Safety of Medisorb® Naltrexone (VIVITROL®)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Bernard Silverman, MD / Vice President, Clinical Development, Alkermes, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK21-003-EXT
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Results first posted 2010-12-08 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — vivitrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medisorb naltrexone 380 mg (Experimental): Intramuscular (IM) injection administered once every 4 weeks for up to 48 weeks.
  Interventions: Drug: Medisorb naltrexone 380 mg
- Medisorb naltrexone 190 mg (Experimental): IM injection administered once every 4 weeks for up to 48 weeks.
  Interventions: Drug: Medisorb naltrexone 190 mg

INTERVENTIONS:
Drug: Medisorb naltrexone 190 mg — naltrexone for extended-release injectable suspension
  Arms: Medisorb naltrexone 190 mg
Drug: Medisorb naltrexone 380 mg — naltrexone for extended-release injectable suspension
  Other Names: VIVITROL
  Arms: Medisorb naltrexone 380 mg

SUMMARY:
This was a Phase 3 multicenter extension of Alkermes' Study ALK21-003 (NCT01218958 [the base study]) that evaluated the safety of Medisorb® naltrexone (VIVITROL®) administered every 4 weeks for 48 weeks (13 injections) in alcohol-dependent adults who had completed Study ALK21-003.

DETAILED DESCRIPTION:
All participants in this study received Medisorb naltrexone at double-blinded dose strengths (ie, 190 mg or 380 mg); no participant received placebo. Participants who had received Medisorb naltrexone in Study ALK21-003 (NCT01218958) continued to receive the same dose strength in this extension study. Those who had received placebo for Medisorb naltrexone 190 mg in the base study were given Medisorb naltrexone 190 mg. Participants who had received placebo for Medisorb naltrexone 380 mg in the base study were given Medisorb naltrexone 380 mg.

Neither the identity or dose of the treatment received in the base study, nor the Medisorb naltrexone dose strength (190 mg or 380 mg) received in this extension were revealed to any participant, the investigator, or any blinded member of the clinical study team during the conduct of the base study or this extension.

All participants were encouraged to receive standardized biopsychosocial support at each clinic visit throughout the study; however, unlike the base study, participation was not mandatory.

Participants eligible for this extension study had received all 6 injections of study drug in the base study; those who received Medisorb naltrexone in the base study who also received all 13 injections in this extension therefore had a duration of exposure of approximately 76 weeks (~1.5 years) upon completion of this extension. For participants who had received placebo in the base study, maximum duration of exposure was approx. 48 weeks (1 year).

ELIGIBILITY:
Primary Inclusion Criteria:

* Completed study drug treatment in Study ALK21-003 (base study [NCT01218958])
* Written informed consent for this extension study
* Stable address and telephone; reconfirmation of contact's address and phone
* Women with childbearing potential must agree to continue to use an approved method of birth control throughout study participation

Primary Exclusion Criteria:

* Positive urine drug screen for opioids at Visit 1
* Early termination of study drug in the base study
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2002-08; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L Silverman, MD, Study Director — Alkermes, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medisorb Naltrexone 380 mg | Medisorb Naltrexone 190 mg
Started | 175 | 157
Completed | 71 | 77
Not Completed | 104 | 80

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medisorb Naltrexone 380 mg | Medisorb Naltrexone 190 mg | Total
Number analyzed (Participants) | 175 | 157 | 332
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 168 | 149 | 317
  >=65 years | 7 | 8 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 45.5 (9.6) | 47.4 (10.5) | 46.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 53 | 115
  Male | 113 | 104 | 217
Region of Enrollment [Number; unit: participants]
  United States | 175 | 157 | 332

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting at Least 1 Treatment-emergent Adverse Event (TEAE) While in Study
Description: A TEAE is any adverse event, whether or not considered drug-related, that develops or worsens in severity after study drug administration begins (ie, from the first administration through the end of the follow-up period).
Time Frame: Up to 48 weeks (13 injections), not including base study
Population: All participants who received at least 1 dose of study drug are included in the safety population.
Measure: Number; unit: Participants
Arm/Group | Medisorb Naltrexone 380 mg | Medisorb Naltrexone 190 mg
Number analyzed (Participants) | 175 | 157
Participants | 143 | 130

ADVERSE EVENTS:
Time Frame: 1 year (Baseline to Week 52)
Groups:
- Medisorb Naltrexone 380mg--Combined: Includes all participants who received Medisorb naltrexone 380mg in this extension study. Study drug was administered via intramuscular (IM) injection once every 4 weeks.
- Medisorb Naltrexone 190mg--Combined: Includes all participants who received Medisorb naltrexone 190mg in this extension study. Study drug was administered via intramuscular (IM) injection once every 4 weeks.
- Placebo to 380mg: Includes participants who received placebo in the base study but switched to Medisorb naltrexone 380mg in this extension. Study drug was administered via intramuscular (IM) injection once every 4 weeks.
- 380mg to 380mg: Includes participants who received Medisorb naltrexone 380mg in the base study and continued with the same dose strength in this extension. Study drug was administered via intramuscular (IM) injection once every 4 weeks.
- Placebo to 190mg: Includes participants who received placebo in the base study but switched to Medisorb naltrexone 190mg in this extension. Study drug was administered via intramuscular (IM) injection once every 4 weeks.
- 190mg to 190mg: includes participants who received Medisorb naltrexone 190mg in the base study and continued with the same dose strength in this extension. Study drug was administered via intramuscular (IM) injection once every 4 weeks.
Arm/Group | Medisorb Naltrexone 380mg--Combined | Medisorb Naltrexone 190mg--Combined | Placebo to 380mg | 380mg to 380mg | Placebo to 190mg | 190mg to 190mg
Serious Adverse Events (participants affected / at risk) | 6/175 | 12/157 | 2/60 | 4/115 | 2/55 | 10/102
Other Adverse Events (participants affected / at risk) | 143/175 | 130/157 | 51/60 | 92/115 | 46/55 | 84/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 380mg--Combined (N=175) | Medisorb Naltrexone 190mg--Combined (N=157) | Placebo to 380mg (N=60) | 380mg to 380mg (N=115) | Placebo to 190mg (N=55) | 190mg to 190mg (N=102)
Intervertebral disc degeneration NOS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Drug abuser NOS (Social circumstances) | 1 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cholecystitis acute NOS (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Limb injury NOS (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pancreatic carcinoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 3 | 0 | 0 | 2 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 380mg--Combined (N=175) | Medisorb Naltrexone 190mg--Combined (N=157) | Placebo to 380mg (N=60) | 380mg to 380mg (N=115) | Placebo to 190mg (N=55) | 190mg to 190mg (N=102)
Nasopharyngitis (Infections and infestations) | 16 | 21 | 8 | 8 | 6 | 15
Upper respiratory tract infection NOS (Infections and infestations) | 18 | 18 | 6 | 12 | 7 | 11
Sinusitis NOS (Infections and infestations) | 7 | 9 | 5 | 2 | 4 | 5
Influenza (Infections and infestations) | 11 | 1 | 4 | 7 | 0 | 1
Bronchitis NOS (Infections and infestations) | 6 | 3 | 3 | 3 | 0 | 3
Gastroenteritis viral NOS (Infections and infestations) | 7 | 1 | 1 | 6 | 0 | 1
Injection site induration (General disorders) | 11 | 5 | 9 | 2 | 4 | 1
Fatigue (General disorders) | 15 | 10 | 8 | 7 | 5 | 5
Injection site pain (General disorders) | 10 | 8 | 4 | 6 | 6 | 2
Influenza like illness (General disorders) | 3 | 12 | 2 | 1 | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 9 | 6 | 10 | 5 | 4
Pain in limb (Musculoskeletal and connective tissue disorders) | 10 | 5 | 5 | 5 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 9 | 2 | 9 | 2 | 7
Nausea (Gastrointestinal disorders) | 17 | 14 | 6 | 11 | 10 | 4
Vomiting NOS (Gastrointestinal disorders) | 5 | 8 | 3 | 2 | 1 | 7
Insomnia (Psychiatric disorders) | 11 | 11 | 4 | 7 | 4 | 7
Depression (Psychiatric disorders) | 5 | 15 | 3 | 2 | 8 | 7
Anxiety NEC (Psychiatric disorders) | 5 | 4 | 2 | 3 | 3 | 1
Alcoholism (Psychiatric disorders) | 2 | 5 | 0 | 2 | 4 | 1
Headache NOS (Nervous system disorders) | 18 | 20 | 8 | 10 | 4 | 16
Dizziness (Nervous system disorders) | 4 | 7 | 1 | 3 | 4 | 3
Back injury NOS (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 1 | 3 | 0
Rash NOS (Skin and subcutaneous tissue disorders) | 4 | 4 | 3 | 1 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 1 | 0 | 3
Appetite decreased NOS (Metabolism and nutrition disorders) | 4 | 4 | 2 | 2 | 4 | 0
Seasonal allergy (Immune system disorders) | 1 | 4 | 1 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should a PI wish to disclose results, the Sponsor will review the results communications prior to public release and can embargo results communications for a period of at least 30 days prior to the submission, for review and approval. Revisions will be negotiated in good faith by the Investigator and Sponsor and may be submitted for publication or disclosed by the Investigator only following receipt of written approval from the Sponsor.